CLINICAL TRIAL: NCT03348683
Title: Propranolol Versus Placebo for Induction of Labor in Nulliparous Patients: a Double-blind Randomized Controlled Trial
Brief Title: Propranolol Versus Placebo for Induction of Labor in Nulliparous Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, joanne stone, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 17-1441
Record Dates: First submitted 2017-11-10; First posted 2017-11-21 (Actual); Results first posted 2019-12-26 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: Induction; Labor; Propranolol
MeSH Terms: interventions — Propranolol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study drug and placebo will be randomized and mixed to appear identical by the Mount Sinai Investigational Drug Service (IDS). The randomization code will be kept by the lead pharmacist of the IDS until completion of the trial, at which point data will be unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Propranolol (Experimental): 2mg of IV push
  Interventions: Drug: Propranolol
- Placebo (Placebo Comparator): an equivalent quantity in milliliters of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — After induction is started with Foley or misoprostol placement, 30 minutes will pass before administration of the one-time study medication, IV Propanolol.
  Arms: Propranolol
Drug: Placebo — After induction is started with Foley or misoprostol placement, 30 minutes will pass before administration of IV Saline
  Other Names: saline
  Arms: Placebo

SUMMARY:
A randomized, prospective trial will be offered to women admitted to the labor floors at Mount Sinai Medical Center for labor induction.

DETAILED DESCRIPTION:
Induction of labor is a common obstetric procedure, which is performed to provoke the onset of labor and lead to delivery of the fetus. While some early studies suggested a possible increased rate of cesarean with induction of labor, more recent meta-analyses have shown that induction does not influence this rate. There is data from small randomized studies that demonstrates the effectiveness of propranolol, a non-selective beta-blocker, for induction of labor. This literature suggests a decrease in the amount of time to delivery and a possible reduction in cesarean section rates when propranolol is used in conjunction with oxytocin for induction of labor compared to oxytocin alone.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women undergoing induction of labor
* >37 weeks' gestational age
* Non-anomalous, singleton cephalic presenting fetus.

Exclusion Criteria:

* Multiple gestations, known fetal anomalies
* Maternal cardiac or hypertensive disease
* Chronic beta blocker use
* Bronchial asthma
* Maternal or fetal indication for immediate delivery.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant patients are the only subjects eligible for study
Enrollment: 240 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Stone, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BLACK JW, CROWTHER AF, SHANKS RG, SMITH LH, DORNHORST AC. A NEW ADRENERGIC BETARECEPTOR ANTAGONIST. Lancet. 1964 May 16;1(7342):1080-1. doi: 10.1016/s0140-6736(64)91275-9. No abstract available. PMID 14132613
- [Background] Moghadam AD, Jaafarpour M, Khani A. Comparison effect of oral propranolol and oxytocin versus oxytocin only on induction of labour in nulliparous women (a double blind randomized trial). J Clin Diagn Res. 2013 Nov;7(11):2567-9. doi: 10.7860/JCDR/2013/5704.3613. Epub 2013 Nov 10. PMID 24392402
- [Background] Kashanian M, Fekrat M, Zarrin Z, Ansari NS. A comparison between the effect of oxytocin only and oxytocin plus propranolol on the labor (a double blind randomized trial). J Obstet Gynaecol Res. 2008 Jun;34(3):354-8. doi: 10.1111/j.1447-0756.2008.00790.x. PMID 18588611
- [Background] Pergialiotis V, Frountzas M, Prodromidou A, Prapa S, Perrea DN, Vlachos GD. Propranolol and oxytocin versus oxytocin alone for induction and augmentation of labor: a meta-analysis of randomized trials. Arch Gynecol Obstet. 2016 Apr;293(4):721-9. doi: 10.1007/s00404-015-3991-8. Epub 2015 Dec 22. PMID 26695642
- [Background] Pruyn SC, Phelan JP, Buchanan GC. Long-term propranolol therapy in pregnancy: maternal and fetal outcome. Am J Obstet Gynecol. 1979 Oct 15;135(4):485-9. doi: 10.1016/0002-9378(79)90436-8. PMID 573555
- [Background] Sanchez-Ramos L, Quillen MJ, Kaunitz AM. Randomized trial of oxytocin alone and with propranolol in the management of dysfunctional labor. Obstet Gynecol. 1996 Oct;88(4 Pt 1):517-20. doi: 10.1016/0029-7844(96)00223-2. PMID 8841209
- [Background] Ikeda S, Tamaoki H, Akahane M, Nebashi Y. Effects of ritodrine hydrochloride, a beta 2-adrenoceptor stimulant, on uterine motilities in late pregnancy. Jpn J Pharmacol. 1984 Jul;35(3):319-26. doi: 10.1254/jjp.35.319. PMID 6482092
- [Background] Meidahl Petersen K, Jimenez-Solem E, Andersen JT, Petersen M, Brodbaek K, Kober L, Torp-Pedersen C, Poulsen HE. beta-Blocker treatment during pregnancy and adverse pregnancy outcomes: a nationwide population-based cohort study. BMJ Open. 2012 Jul 19;2(4):e001185. doi: 10.1136/bmjopen-2012-001185. Print 2012. PMID 22815467
- [Background] Omar HA, Rhodes LA, Ramirez R, Arsich J, Einzig S. Alteration of human placental vascular tone by antiarrhythmic medications in vitro. J Cardiovasc Electrophysiol. 1996 Dec;7(12):1197-203. doi: 10.1111/j.1540-8167.1996.tb00498.x. PMID 8985808
- [Background] Palomaki O, Uotila J, Tammela O, Kaila T, Lavapuro M, Huhtala H, Tuimala R. A double blind, randomized trial on augmentation of labour with a combination of intravenous propranolol and oxytocin versus oxytocin only. Eur J Obstet Gynecol Reprod Biol. 2006 Mar 1;125(1):44-9. doi: 10.1016/j.ejogrb.2005.06.016. Epub 2005 Jul 26. PMID 16051416
- [Derived] Bigelow CA, Pan S, Overbey JR, Stone J. Propranolol for Induction of Labor in Nulliparas trial a double-blind, randomized, placebo-controlled trial. Am J Obstet Gynecol MFM. 2021 Mar;3(2):100301. doi: 10.1016/j.ajogmf.2020.100301. Epub 2021 Jan 6. PMID 33421647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First enrollment 12-11-2017, final enrollment 12/11/2018. Enrollment occurred on the labor floor of the Mount Sinai Hospital.
Groups:
- Propranolol: After induction was started with Foley or misoprostol placement, 30 minutes passed before administration of propranolol 2mg of IV push
- Placebo: After induction was started with Foley or misoprostol placement, 30 minutes passed before administration of an equivalent quantity in milliliters of IV normal saline
Period: Overall Study
Arm/Group | Propranolol | Placebo
Started | 121 | 119
Completed | 121 | 119
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo | Total
Number analyzed (Participants) | 121 | 119 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.70 (5.72) | 31.61 (6.37) | 31.66 (6.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 119 | 240
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 5 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 11 | 27
  White | 72 | 83 | 155
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 17 | 20 | 37
Body Mass Index (BMI) at admission [Mean (Standard Deviation); unit: kg/m^2] | 29.04 (5.34) | 28.89 (4.40) | 28.97 (4.89)
Gestational Age (GA) at admission [Median (Inter-Quartile Range); unit: months] | 39.7 [39 to 40.9] | 40.1 [39.3 to 40.9] | 40.0 [39.1 to 40.9]
Married [Count of Participants; unit: Participants] | 94 | 97 | 191
Private Insurance [Count of Participants; unit: Participants] | 101 | 93 | 194
In vitro Fertilization (IVF) [Count of Participants; unit: Participants] | 18 | 19 | 37
Fetal Growth Restriction [Count of Participants; unit: Participants] | 8 | 3 | 11
Tobacco Use [Count of Participants; unit: Participants] | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time From Beginning of Induction to Delivery
Description: The time of induction (based on time of foley balloon placement for cervical ripening or misoprostol administration) to the time of delivery of the infant.
Time Frame: average of 24 hours
Population: N=154 - only those who delivered vaginally
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 75 | 79
hours | 13.8 (5.4) | 14.3 (5.3)

2. Secondary Outcome: Number of Participants With Various Mode of Delivery
Description: Number of various mode of delivery - count of Vaginal delivery, vacuum assisted vaginal delivery, forceps assisted vaginal delivery, cesarean section
Time Frame: average of 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 121 | 119
Participants
  Spontaneous vaginal delivery | 64 | 61
  Vacuum assisted vaginal delivery | 3 | 10
  Forceps assisted vaginal delivery | 8 | 8
  Cesarean section | 46 | 40

3. Secondary Outcome: Duration of Latent
Description: Time of latent labor defined as <6cm of cervical dilation.
Time Frame: average of 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 121 | 119
hours | 11.0 (5.0) | 11.2 (4.5)

4. Secondary Outcome: Number of Participants With Maternal Morbidity Composite Score = 1
Description: Composite maternal morbidity score consists of a count of postpartum hemorrhage, transfusion, hysterectomy, placental abruption, chorioamnionitis, shoulder dystocia, episiotomy, higher order laceration, and ICU admission.
  The composite score was computed as a score of 1 for any indication of maternal morbidity, that is the participant experienced at least one maternal morbidity, and the components are given equal weights. Participants who had no evidence of the predefined maternal morbidities are subsequently given a score of 0. The minimum is 0 and maximum is 1.
Time Frame: average of 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 121 | 119
Participants | 35 | 49

5. Secondary Outcome: Number of Participants With Postpartum Hemorrhage
Description: Greater than 500cc of blood expelled during a vaginal delivery or greater than 1000cc of blood expelled during a cesarean section
Time Frame: 30 minutes from drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 121 | 119
Participants | 15 | 26

6. Secondary Outcome: Number of Fetus With Heart Rate Decelerations
Description: Count of fetus with fetal heart rate decelerations within 30 minutes of study drug administration
Time Frame: 30 minutes from drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 121 | 119
Participants | 15 | 13

7. Secondary Outcome: Number of Fetus With Fetal Bradycardia
Description: Count of fetus with fetal bradycardia (<110bpm for >10 minutes within 30 minutes of study drug administration)
Time Frame: 30 minutes from drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 121 | 119
Participants | 1 | 0

8. Secondary Outcome: Number of Neonates With Neonatal Outcome Composite Score = 1
Description: Composite neonatal outcome score was for any of the following morbidity: Neonatal Intensive Care Unit (NICU) admission, respiratory support (CPAP, nasal cannula, intubation), culture proven sepsis, radiographically proven intracranial hemorrhage, necrotizing enterocolitis, hypoglycemia (for those infants who had sugar checked), and neonatal death.
  The composite score was computed as a score of 1 for any indication of neonatal morbidity - neonates who experienced at least one morbidity and the components are given equal weights. Patients who had no evidence of the predefined neonatal morbidities are subsequently given a score of 0. The minimum is 0 and maximum is 1.
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 121 | 119
Participants | 21 | 28

9. Secondary Outcome: Number of Neonates With Hypoglycemia
Description: Neonatal outcome - Number of neonates with hypoglycemia (blood glucose <50).
  This population includes only the neonates who had heelsticks to check their blood glucose, which is not a universal practice and was not required by the protocol or IRB. The neonates included were those who met the nursery's risk-based protocol to check blood glucose after birth (ex: infants of diabetic mothers, fetal growth restriction, macrosomia, or symptoms suggestive of hypoglycemia)
Time Frame: Day 1
Population: This population includes the neonates who had heelsticks to check their blood glucose.
Measure: Count of Participants; unit: Participants
Arm/Group | Propranolol | Placebo
Number analyzed (Participants) | 45 | 49
Participants | 11 | 8

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Propranolol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/119
Serious Adverse Events (participants affected / at risk) | 1/121 | 0/119
Other Adverse Events (participants affected / at risk) | 16/121 | 13/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Propranolol (N=121) | Placebo (N=119)
Fetal bradycardia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Fetal bradycardia within 30 minutes of study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Propranolol (N=121) | Placebo (N=119)
Maternal hypotension (Vascular disorders) | 1 | 0 — Maternal hypotension <80/40 within 30 minutes of study drug (no pressors required)
Fetal heart rate decelerations (Pregnancy, puerperium and perinatal conditions) | 15 | 13 — Fetal heart rate decelerations within 30 minutes of study drug

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT03348683/Prot_SAP_000.pdf